CLINICAL TRIAL: NCT00106392
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess the Safety and Efficacy of Prograf (Tacrolimus, FK 506) for the Prevention of Erectile Dysfunction Following Bilateral Nerve-sparing Radical Prostatectomy
Brief Title: A Safety and Efficacy Study of Prograf in the Prevention of Erectile Dysfunction After Radical Prostatectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sr Manager Clinical Trial Registries, Astellas Pharma US, Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20-03-001
Record Dates: First submitted 2005-03-23; First posted 2005-03-24 (Estimated); Results first posted 2010-10-28 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-11

CONDITIONS: Erectile Dysfunction; Prostate Cancer
Keywords: Treatment effectiveness; Treatment efficacy; Investigational, Therapies; Immunosuppressant; Erectile dysfunction; Prostatectomy
MeSH Terms: conditions — Erectile Dysfunction; Prostatic Neoplasms | interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tacrolimus (Experimental): Preoperatively: Tacrolimus 2 mg oral daily from 4 to 10 days prior to surgery through hospital discharge; Postoperatively: Tacrolimus 3 mg oral daily at time of hospital discharge through 6 months of follow up.
  Interventions: Drug: Tacrolimus
- Placebo (Placebo Comparator): Preoperatively: Matching placebo oral daily from 4 to 10 days prior to surgery through hospital discharge; Postoperatively: Matching placebo oral daily at time of hospital discharge through 6 months of follow up.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tacrolimus — oral
  Other Names: Prograf, FK506
  Arms: Tacrolimus
Drug: Placebo — oral
  Arms: Placebo

SUMMARY:
The purpose of the study is to compare the safety and effectiveness of Prograf in the prevention of erectile dysfunction in men after a radical prostatectomy.

DETAILED DESCRIPTION:
The purpose of the study is to compare the safety and efficacy of Prograf versus placebo in the prevention of erectile dysfunction in men after a bilateral nerve-sparing radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Male scheduled to undergo bilateral nerve sparing radical prostatectomy for prostate cancer.

Exclusion Criteria:

* Patient is > 65 years of age
* Patient has been diagnosed with Type 1 or Type 2 diabetes
* Patient is actively smoking on a daily basis

Max Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2005-02; Primary Completion 2008-04 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma US, Inc.
Locations (5):
- United States (5):
  - Ann Arbor, Michigan
  - New York, New York
  - Cleveland, Ohio
  - Nashville, Tennessee
  - Houston, Texas

REFERENCES:
- [Derived] Mulhall JP, Klein EA, Slawin K, Henning AK, Scardino PT. A Randomized, Double-Blind, Placebo-Controlled Trial to Assess the Utility of Tacrolimus (FK506) for the Prevention of Erectile Dysfunction Following Bilateral Nerve-Sparing Radical Prostatectomy. J Sex Med. 2018 Sep;15(9):1293-1299. doi: 10.1016/j.jsxm.2018.07.009. PMID 30224019
- See also: Link to prescribing information — http://www.astellas.us/docs/prograf.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tacrolimus | Placebo
Started | 62 | 69
Baseline Participants | 59 (3 patients withdrew: 2 prior to surgery and study drug; 1 took study drug but did not have surgery) | 65 (4 patients withdrew: all prior to surgery and study drug)
Full Analysis Set (FAS) | 53 | 61
Completed | 36 | 42
Not Completed | 26 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tacrolimus | Placebo | Total
Number analyzed (Participants) | 59 | 65 | 124
Age Continuous [Mean (Standard Deviation); unit: years] | 55.1 (6.2) | 54.1 (6.2) | 54.6 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 59 | 65 | 124
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaskan Native | 0 | 1 | 1
  Black or African American | 4 | 1 | 5
  White | 55 | 63 | 118

OUTCOME MEASURES:

1. Primary Outcome: Erectile Function Domain Score Between Treated and Untreated Groups
Description: Erectile function was assessed using the International Index of Erectile Function (IIEF) questionnaire, which consists of 15 questions. The erectile function domain score is calculated as a sum of scores from questions 1-5 and 15. A clinically meaningful difference is 5 points. The scores range from 1 to 30 points where a higher score indicates better erectile function. Normal erectile function is defined as greater than or equal to 24 points.
Time Frame: 18 months
Population: The number of participants analyzed represents Full Analysis Set (FAS), which is defined as participants evaluated for Efficacy and Safety.
  Only participants with complete IIEF questionnaire data at 18 months are included in the calculation.
Measure: Median (Full Range); unit: Erectile Function Domain Score
Arm/Group | Tacrolimus | Placebo
Number analyzed (Participants) | 32 | 38
Erectile Function Domain Score | 18.0 [1.0 to 30.0] | 23.5 [4.0 to 30.0]
Statistical Analysis 1: Comparison: Tacrolimus vs Placebo; A group sequential design using the O'Brien and Fleming stopping rule will require 58 evaluable patients per group to detect a 5-point difference in the Erectile Function domain of the IIEF with a power of 80% and an overall significance level of 5%; Test type: Superiority or Other; p = 0.111, Wilcoxon (Mann-Whitney) — P-Values were not adjusted

2. Secondary Outcome: Percentage of Patients Achieving Normal Spontaneous Erectile Function as Measured by the Erectile Function (EF) Domain Score
Description: Erectile function was assessed using the International Index of Erectile Function (IIEF) questionnaire, which consists of 15 questions. The erectile function domain score is calculated as a sum of scores from questions 1-5 and 15. A clinically meaningful difference is 5 points. The scores range from 1 to 30 points where a higher score indicates better erectile function. Normal erectile function is defined as greater than or equal to 24 points.
  Percentages represent the proportions of participants who achieved normal erectile function at any time during the 24 months.
Time Frame: 24 months
Population: The number of participants analyzed represents Full Analysis Set (FAS), which is defined as participants evaluated for Efficacy and Safety.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tacrolimus | Placebo
Number analyzed (Participants) | 53 | 61
Percentage of Participants | 45.3 | 54.1
Statistical Analysis 1: Comparison: Tacrolimus vs Placebo; Test type: Superiority or Other; p = 0.453, Fisher Exact

3. Secondary Outcome: Time Taken to Achieve Normalization of the Erectile Function (EF) Domain Score
Description: Erectile function was assessed using the International Index of Erectile Function (IIEF) questionnaire, which consists of 15 questions. The EF domain score is calculated as a sum of scores from questions 1-5 and 15. A clinically meaningful difference is 5 points. Scores range from 1-30 points where a higher score indicates better erectile function. Normal erectile function is defined as greater than or equal to 24 points.Time to achieve normalization of the EF domain score was calculated based on the date of the assessment during which the EF domain score was first greater than or equal to 24.
Time Frame: 24 months
Population: The number of participants analyzed represents Full Analysis Set (FAS), which is defined as participants evaluated for Efficacy and Safety.
  Only participants who achieved normal erectile function are included in the calculation.
Measure: Median (Full Range); unit: Days
Arm/Group | Tacrolimus | Placebo
Number analyzed (Participants) | 24 | 33
Days | 104.5 [28.0 to 753.0] | 180.0 [29.0 to 730.0]
Statistical Analysis 1: Comparison: Tacrolimus vs Placebo; Test type: Superiority or Other; p = 0.790, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Percentage of Patients Considered Successful Responders to Impotence Medications
Description: Patients were identified as successful responders if they answered affirmatively in the Patient Sexual Encounter Diary regarding successful sexual intercourse after using impotence medication.
Time Frame: 24 months
Population: The number of participants analyzed represents Full Analysis Set (FAS), which is defined as participants evaluated for Efficacy and Safety.
  Only participants who used any impotence medications were included in the calculation.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tacrolimus | Placebo
Number analyzed (Participants) | 52 | 58
Percentage of Participants | 73.1 | 86.2
Statistical Analysis 1: Comparison: Tacrolimus vs Placebo; Test type: Superiority or Other; p = 0.099, Fisher Exact

5. Secondary Outcome: Time to Achieve Response to Impotence Medications
Description: Time to achieve response to impotence medication was calculated based on the date of the assessment during which the first successful response was recorded. The specific date of the actual response is not reflected; only that it occurred since the previous study visit.
Time Frame: 24 months
Population: The number of participants analyzed represents Full Analysis Set (FAS), which is defined as participants evaluated for Efficacy and Safety.
  Only participants who had a successful response to impotence medications were included in the calculations.
Measure: Median (Full Range); unit: Days
Arm/Group | Tacrolimus | Placebo
Number analyzed (Participants) | 38 | 50
Days | 102.0 [34.0 to 730.0] | 113.5 [29.0 to 821.0]
Statistical Analysis 1: Comparison: Tacrolimus vs Placebo; Test type: Superiority or Other; p = 0.575, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Continence Level as Quantified by Part I of the Prostate Health-Related Quality of Life Questionnaire
Description: Part 1 Urinary Function- Prostate Health-Related Quality-of-Life (QOL) Questionnaire consists of 16 questions asking patients about their continence and urinary habits over the previous four weeks. The responses to all 16 of these questions were added together to calculate an overall score for urinary function. The minimum possible score is 16 and the maximum possible score is 79. A higher score indicates a lower continence level.
Time Frame: 24 months
Population: The number of participants analyzed represents Full Analysis Set (FAS), which is defined as participants evaluated for Efficacy and Safety.
  Only participants with a Prostate Health-Related QOL questionnaire at 24 months were included in the calculation.
Measure: Median (Full Range); unit: Overall Score of Urinary Function
Arm/Group | Tacrolimus | Placebo
Number analyzed (Participants) | 39 | 47
Overall Score of Urinary Function | 22.0 [16.0 to 49.0] | 22.0 [16.0 to 52.0]
Statistical Analysis 1: Comparison: Tacrolimus vs Placebo; Test type: Superiority or Other; p = 0.879, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: SAEs and AEs as defined below were collected through month 6.
Description: Serious Adverse Events possibly related to study drug were collected.
  The only other Adverse Events collected were those associated with study drug dose changes.
  Subjects who experienced an Adverse Event with the same preferred term multiple times were only counted once.
Arm/Group | Tacrolimus | Placebo
Serious Adverse Events (participants affected / at risk) | 1/59 | 0/65
Other Adverse Events (participants affected / at risk) | 7/59 | 5/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus (N=59) | Placebo (N=65)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus (N=59) | Placebo (N=65)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 2
Renal disorder (Renal and urinary disorders) | 3 | 3

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose, and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript at least 30 days prior to publication to ensure that no confidential information of Sponsor is included in the document.